CLINICAL TRIAL: NCT02943590
Title: STOP-CA (Statins TO Prevent the Cardiotoxicity From Anthracyclines)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Tomas G. Neilan, MD, MD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-440
Record Dates: First submitted 2016-10-21; First posted 2016-10-24 (Estimated); Results first posted 2023-12-18 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure
Keywords: Cancer Treatment Related to Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo will be administered at a pre determined dose The drug is taken by mouth, once a day (evening)
  Interventions: Drug: Placebo
- Atorvastatin (Experimental): Atorvastatin will be administered at a pre determined dose The drug is taken by mouth, once a day (evening)
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Placebo — A pill taken once a day
  Arms: Placebo
Drug: Atorvastatin — A pill taken once a day
  Other Names: Lipitor
  Arms: Atorvastatin

SUMMARY:
This research study will test whether atorvastatin, a drug commonly prescribed for reducing cholesterol levels, can protect the heart during chemotherapy with doxorubicin. Atorvastatin is from a family of medications that are commonly called "statins"

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the effectiveness of a drug and determine whether the investigational drug works in treating a specific disease. "Investigational" means that the drug is being studied.

The chemotherapy drug that the participant have been scheduled to be treated with, Doxorubicin, has been associated with the development of heart failure in some patients.

This research study is testing whether Atorvastatin can protect the hearts of patients being treated with Doxorubicin and can reduce cardiac injury and the risk of heart failure. Atorvastatin is not approved by the FDA (the U.S. Food and Drug Administration) for use to reduce the cardiac injury after Doxorubicin. Atorvastatin is approved by the FDA for lowering cholesterol and for reducing the risk of heart attack and stroke. The heart is a muscle that pumps blood and Atorvastatin may protect the heart by preserving cardiac muscle function.

The investigators will test whether atorvastatin protects the heart using a combination of imaging tests on the participants heart, blood tests, and stress testing. The imaging tests will involve an echocardiogram (an echo) and cardiac magnetic resonance (CMR), a type of magnetic resonance imaging (MRI) scan.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* All patients with newly diagnosed NHL and HL
* Scheduled to receive anthracycline-based therapy

Exclusion Criteria:

* Statin use or Statin use is indicated based on guidelines
* Pregnancy or breastfeeding
* Unable to provide informed consent
* Unexplained persistent elevation of transaminases (>3 times upper limits of normal)
* Concomitant use of cyclosporine
* Renal failure: estimated glomerular filtration <45 mL/min/1.73 m2
* Contraindication to a CMR (metallic object, severe claustrophobia, pacemaker, vascular clip
* LVEF of <50% at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2023-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tomas G Neilan, MD, Principal Investigator — Massachusetts General Hospital
Locations (4):
- United States (3):
  - Massachusetts general Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Pennsylvania Medical System, Philadelphia, Pennsylvania
- McGill University Health Center, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Juhasz V, Drobni ZD, Quinaglia T, Gilman HK, Brendel JM, Suero-Abreu GA, Ghamari A, Heemelaar JC, Neuberg DS, Han Y, Ky B, Kwong RY, Januzzi JL, Asnani A, Mousavi N, Redd RA, Jerosch-Herold M, Scherrer-Crosbie M, Neilan TG. Atorvastatin and Aortic Stiffness During Anthracycline-Based Chemotherapy: A Secondary Analysis of a Randomized Clinical Trial. JAMA Cardiol. 2026 Jan 1;11(1):68-76. doi: 10.1001/jamacardio.2025.4548. PMID 41205202
- [Derived] Juhasz V, Drobni ZD, Quinaglia T, Gilman HK, Suero-Abreu GA, Ghamari A, Heemelaar JC, Neuberg DS, Han Y, Ky B, Kwong RY, Januzzi JL, Asnani A, Mousavi N, Redd RA, Jerosch-Herold M, Scherrer-Crosbie M, Neilan TG. Atorvastatin and left atrial function during anthracycline-based chemotherapy. J Cardiovasc Magn Reson. 2025 Winter;27(2):101946. doi: 10.1016/j.jocmr.2025.101946. Epub 2025 Aug 26. PMID 40876541
- [Derived] Juhasz V, Quinaglia T, Drobni ZD, Heemelaar JC, Neuberg DS, Han Y, Ky B, Kwong RY, Januzzi JL, Asnani A, Redd RA, Mousavi N, Jerosch-Herold M, Scherrer-Crosbie M, Neilan TG. Atorvastatin and Myocardial Extracellular Volume Expansion During Anthracycline-Based Chemotherapy. JACC CardioOncol. 2025 Feb;7(2):125-137. doi: 10.1016/j.jaccao.2024.11.008. Epub 2025 Jan 28. PMID 39967198
- [Derived] Neilan TG, Quinaglia T, Onoue T, Mahmood SS, Drobni ZD, Gilman HK, Smith A, Heemelaar JC, Brahmbhatt P, Ho JS, Sama S, Svoboda J, Neuberg DS, Abramson JS, Hochberg EP, Barnes JA, Armand P, Jacobsen ED, Jacobson CA, Kim AI, Soumerai JD, Han Y, Friedman RS, Lacasce AS, Ky B, Landsburg D, Nasta S, Kwong RY, Jerosch-Herold M, Redd RA, Hua L, Januzzi JL, Asnani A, Mousavi N, Scherrer-Crosbie M. Atorvastatin for Anthracycline-Associated Cardiac Dysfunction: The STOP-CA Randomized Clinical Trial. JAMA. 2023 Aug 8;330(6):528-536. doi: 10.1001/jama.2023.11887. PMID 37552303

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1:1 randomization
Period: Overall Study
Arm/Group | Placebo | Atorvastatin
Started | 150 | 150
Completed | 144 | 142
Not Completed | 6 | 8

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo group
- Atorvastatin: Atorvastatin group
- Total: Total of all reporting groups
Arm/Group | Placebo | Atorvastatin | Total
Number analyzed (Participants) | 150 | 150 | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 130 | 130 | 260
  >=65 years | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (16) | 50 (17) | 50 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 68 | 142
  Male | 76 | 82 | 158
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 4 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 131 | 135 | 266
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 6 | 14
Region of Enrollment [Number; unit: participants]
  Canada | 10 | 10 | 20
  United States | 140 | 140 | 280
LVEF [Mean (Standard Deviation); unit: %] | 62.5 (4.9) | 63 (4.5) | 63 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Individuals in Each Group With a Significant Decline in the LVEF.
Description: To determine if the administration of statins is associated with a lower percentage of individuals who experience a significant decline in the LVEF at 12 months. The primary outcome was the percentage of participants with an absolute decline in left ventricular ejection fraction (LVEF) of>10% from prior to chemotherapy to a final value of <55% over 12 months.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Atorvastatin
Number analyzed (Participants) | 144 | 142
Participants | 22 | 9

2. Secondary Outcome: The Percentage of Participants in Each Group With New Onset Heart Failure.
Description: To determine whether statins reduce the percentage of participants in each group with new onset heart failure after anthracyclines.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Atorvastatin
Number analyzed (Participants) | 144 | 142
Participants | 6 | 3

3. Secondary Outcome: Myocardial Extracellular Volume by Cardiac MRI.
Description: The myocardial extracellular volume (ECV) is the proportion of the myocardium that is estimated to be of extracellular space. Myocardium consists of intracellular space and extracellular space. This measure is an imaging estimate of the extracellular space. The extracellular space can be expanded in diseases where myocardial fibrosis is increased. Thus, this measure is often used as an estimate for the proportion of fibrosis in the heart. It can be expressed as a percentage. Here, based on published literature, we used a cut off of a 3% increase in the ECV from baseline to follow-up as a meaningful increase and compared the propositions of persons with that 3% increase in each group. We are comparing the proportion of persons in each group with a 3% or greater increase in the ECV.
Time Frame: 1 Year
Population: Persons with available and high quality MRI data where the variable could be measured.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Atorvastatin
Number analyzed (Participants) | 62 | 65
Participants | 29 | 8

4. Secondary Outcome: Global Longitudinal Strain (GLS)
Description: GLS is a sensitive measure of cardiac systolic function. Anthracyclines can be associated with impaired global longitudinal strain (GLS). Whether atorvastatin protects against a decline in LV GLS is unknown. GLS is expressed as a percentage. A ≥15% relative decrease in LV GLS was used as a cut off for a significant decrease in GLS based on published data. The Proportions of participants with a relative reduction of ≥15% in LV GLS were evaluated in each group.
Time Frame: 1 year
Population: The number of persons in each group with high quality imaging data where the variable could be analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Those in the placebo group
- Statin: Those randomized to atorvastatin
Arm/Group | Placebo | Statin
Number analyzed (Participants) | 90 | 98
Participants | 28 | 19

ADVERSE EVENTS:
Time Frame: 12 months
Description: No difference
Arm/Group | Placebo | Atorvastatin
All-Cause Mortality (participants affected / at risk) | 4/150 | 4/150
Serious Adverse Events (participants affected / at risk) | 0/150 | 0/150
Other Adverse Events (participants affected / at risk) | 21/150 | 28/150
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=150) | Atorvastatin (N=150)
Muscle pain (Musculoskeletal and connective tissue disorders) | 21 | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2017-02-02): https://cdn.clinicaltrials.gov/large-docs/90/NCT02943590/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-07): https://cdn.clinicaltrials.gov/large-docs/90/NCT02943590/SAP_001.pdf
  • Informed Consent Form (2022-04-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT02943590/ICF_002.pdf